CLINICAL TRIAL: NCT00300534
Title: Multi-site Study of Rapid Diagnostic Syphilis Assays of Persons Attending STD Clinics in High Syphilis Morbidity Areas
Brief Title: Multi-site Study of Rapid Diagnostic Syphilis Assays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDC-NCHSTP-2875
Record Dates: First submitted 2006-03-02; First posted 2006-03-09 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Syphilis
Keywords: Diagnosis
MeSH Terms: conditions — Syphilis; Disease

ARMS (1):
- Abbott Laboratories Determine test for syphilis (No Intervention): Abbott Laboratories Determine rapid test for syphilis
  Interventions: Device: Abbott Laboratories Determine test for syphilis; Device: Investigational syphilis immunochromatographic strip test

INTERVENTIONS:
Device: Abbott Laboratories Determine test for syphilis
Device: Investigational syphilis immunochromatographic strip test

SUMMARY:
The performance of an investigational immunochromatographic strip (ICS) test for the diagnosis of syphilis is compared with the Abbott Laboratories Determine ICS test. The study population consists of patients with and without syphilis presenting to sexually transmitted disease clinics in five cities in the United States. Specimens include finger-stick whole blood (investigational test only) and whole blood, plasma, and serum by venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients

Exclusion Criteria:

* Less than age 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2002-08; Primary Completion 2005-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Treponema pallidum infection | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Johnson, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (5):
- United States (5):
  - Los Angeles Department of Health Services, Los Angeles, California
  - Fulton County Department of Health, Atlanta, Georgia
  - Chicago Department of Public Health, Chicago, Illinois
  - Bell Flower Clinic, Indianapolis, Indiana
  - New York City Department of Health, New York, New York